

Protocol Version: 2.0 Date: 2020/06/30

NCT Number: NCT0269908

# **Section 5. PROTOCOL**

# **Investigational New Drug (IND)**

PDC-1421 Capsule

(Polygala tenuifolia Willd.)

EDITION NUMBER: Version 2.0
SPONSOR: BioLite, Inc.
RELEASE DATE: 2020/06/30

A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), Part I




# STUDY CONTACT INFORMATION

| SPONSOR | Company: BioLite, Inc. |
|--------------|-------------------------------------------------------|
| | Address: 2F, 20, Sec. 2, Shengyi Rd., Zhubei City, |
| | Hsinchu County, 30261, Taiwan |
| | Phone: +886-3-668-5386 |
| | FAX: +886-3-657-9632 |
| PRINCIPAL | Name: Keith McBurnett, Ph.D. |
| INVESTIGATOR | Title: Professor, Psychiatry, Psychiatry Department, |
| | University of California San Francisco, School of |
| | Medicine |
| | Address: 401 Parnassus Ave., Langley Porter Building, |
| | San Francisco, California, USA |
| | Phone: +1-415-476-7892 |
| CLINICAL | CRO to be retained. |
| MONITOR | |
| STUDY SITE | Hospital: UCSF Medical Center |
| | Address: 401 Parnassus Ave., Langley Porter Building, |
| | San Francisco, California, USA |




# SIGNATURE PAGE

| Study | Title: |
|-------|--------|
|-------|--------|

A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), Part I

I have read this protocol and confirm that to the best of my knowledge it accurately describes the conduct of the study.

#### SPONSOR'S REPRESENTATIVE

| TYPED NAME (S) | TITLE | <u>SIGNATURE</u> | <u>DATE</u> |
|------------------|----------------|------------------|-------------|
| Chi-Hsin R. King | Study Director | | |




# SIGNATURE PAGE

# **Study Title:**

A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), Part I

#### **INVESTIGATOR (S)**

I agree to conduct this clinical study in accordance with the design and specific provisions of this protocol; deviations from the protocol are acceptable only with a mutually agreed upon protocol amendment. I also agree to report all information or data in accordance with the protocol and, in particular, I agree to report any serious adverse experiences as defined in this protocol. I also agree to handle all clinical supplies provided by the Sponsor.

#### **Principal Investigator**

| TYPED NAME (S) | <u>TITLE</u> | <u>SIGNATURE</u> | <u>DATE</u> |
|---|---|---|---|
| Keith McBurnett, Ph.D. | Professor, Psychiatry | | |


# **Table of Contents**

| | Page |
|---|---|
| PROTOCOL SYNOPSIS | 8 |
| LIST OF ABBREVIATIONS/DEFINITIONS | 10 |
| 1. Background Information | 13 |
| 1.1 Description of PDC-1421 Capsule | 13 |
| 1.1.1 Preparation | 13 |
| 1.1.2 Composition | 15 |
| 1.1.3 Storage and Handling | 15 |
| 1.2 Non-clinical Study of PDC-1421 | 15 |
| 1.2.1 Efficacy Pharmacology | 15 |
| 1.2.2 Safety Pharmacology | 19 |
| 1.2.3 Cytochrome P450 Interaction with PDC-1421 | 21 |
| 1.2.4 Toxicology | 21 |
| 1.3 Results of Phase I Clinical Trial Study of PDC-1421 | 23 |
| 1.4 Potential Risk and Benefit | 25 |
| 1.4.1 Potential Risk | 25 |
| 1.4.2 Potential Benefit | 25 |
| 1.4.3 Risk Benefit Ratio | 25 |
| 1.5 Dosage Regimen | 25 |
| 1.6 Compliance with Protocol, Good Clinical Practice (GCP) and Applicable | |
| Requirement | 27 |
| 1.7 Description of the Population to be Studied | 27 |
| 2. Trial Objective | 28 |
| 3. Trial Design. | 28 |
| 3.1 General Design | 28 |
| 3.2 Primary Endpoint | 30 |
| 3.3 Secondary Endpoint | 30 |
| 3.4 Randomization and Blinding | 30 |
| 3.5 Investigational Drug | 30 |
| 3.5.1 Dosage Form and Strength | 30 |
| 3.5.2 Manufacturer | 30 |
| 3.5.3 Route of Administration | 30 |




| 3.5.4 Dosing Regimen, packing and labeling | 31 |
|---|---|
| 3.5.5 Study Drug Storage | 34 |
| 3.6 Premature Termination or Suspension of the Study | 34 |
| 4. Subjects Selection and Withdrawal | 35 |
| 4.1 Inclusion Criteria | 35 |
| 4.2 Exclusion Criteria | 35 |
| 4.3 Subject Recruitment and Screening | 36 |
| 4.4 Subject Identification | 36 |
| 4.4.1 Subject Initial Allocation | 37 |
| 4.4.2 Subject Number Allocation | 37 |
| 4.5 Early Withdrawal of Subjects | 38 |
| 5. Treatment of Subjects | 38 |
| 5.1 Description of Study Drug | 38 |
| 5.2 Treatment Schedule | 38 |
| 5.2.1 Screening Phase (Visit 1) | 39 |
| 5.2.2. Part I Study Treatment Period (Visit 2~8) and Follow-up (Visit 9) | 40 |
| 5.3 Other Medication During the Study | 41 |
| 6. Efficacy Assessments | 42 |
| 6.1 Specification of the efficacy parameters | 42 |
| 6.2 Methods and Timing for Assessing, Recording, and Analyzing of Efficacy | |
| Parameters. | 42 |
| 7. Safety Assessments | 44 |
| 7.1 Specification of Safety Parameters | 44 |
| 7.2 Methods and Timing for Assessing, Recording, and Analyzing of Safety | |
| Parameters | 44 |
| 7.3 Adverse Events (AEs) | 44 |
| 7.4 Serious Adverse Events (SAE) | 45 |
| 7.5 Serious and Unexpected Suspected Adverse Reaction (SUSAR) | 45 |
| 7.6 SAE Report Procedure | 46 |
| 7.6.1 Expedited Reporting of SAEs | 46 |
| 7.6.2 IRB Notification | 46 |
| 7.6.3 Record Retention | 46 |
| 8. Statistic Methods | 47 |
| 8.1 Sample Size Determination | 47 |

#### Confidential



Protocol Number: BLI-1008-001


| 8.2 Statistical Method | 47 |
|--------------------------------------------------------|----|
| 8.3 Analysis of Efficacy and Safety | 47 |
| 8.4 Premature Termination and Handling of Missing Data | 48 |
| 9. Quality Control and Quality Assurance | 49 |
| 9.1 Study Monitoring. | 49 |
| 9.2 Sponsor Auditing | 49 |
| 9.3 Inspected by Regulatory Authorities | 49 |
| 10. Ethical Considerations | 50 |
| 10.1 Confidential | 50 |
| 10.2 Protocol Amendment | 50 |
| 10.3 Informed Consent | 50 |
| 10.4 Institutional Review Board (IRB) | 51 |
| 11. Data Handling and Record Keeping | 52 |
| 11.1 Data Handling and Collection. | 52 |
| 11.1.1 Study Specific Binders | 52 |
| 11.1.2 Responsibilities of Investigators | 52 |
| 11.1.3 Responsibilities of Clinical Monitor | 53 |
| 11.2 Records Retention | 53 |
| 11.2.1 Source Document Retention | 53 |
| 11.2.2 CRF Retention | 54 |
| 11.2.3 Record Maintenance | 54 |
| 11.3 Study Center File Management | 54 |
| 12. Publication Plan | 56 |
| 13. References | 56 |

### Appendix 1

- 1. Form FDA 1572 of Principal-Investigator, Keith McBurnett, Ph.D.
- 2. Curriculum Vitae of Keith McBurnett, Ph.D.

### Appendix 2

Informed Consent Form




# PROTOCOL SYNOPSIS

| Name of sponsor | BioLite, Inc. |
|---|---|
| Name of finished | PDC-1421 Capsule |
| product | |
| Name of active | PDC-1421 |
| ingredient | |
| Protocol title | A Phase II Tolerability and Efficacy Study of PDC-1421 |
| | Treatment in Adult Patients with Attention-Deficit |
| | Hyperactivity Disorder (ADHD), Part I |
| Clinical trial phase | Phase II |
| Study site | Single site |
| Study period | 1 year |
| Study population | Patients with ADHD according to the Diagnosis and |
| | Statistical Manual of Mental Disorders, 5th Edition |
| Primary study | To determine the efficacy profile of PDC-1421 Capsule in |
| objective | ADHD with ADHD Rating Scale-IV (ADHD-RS-IV). |
| Secondary study | To determine the efficacy and safety profile of PDC-1421 |
| objective | Capsule in ADHD with other rating scales. |
| Study design | Part I: open label, dose-escalating study |
| Sample size | Maximum 6 subjects |
| Test product | PDC-1421 Capsule |
| Dose and regimen | 1 and 2 capsules thrice daily, p.o., after meal |
| <b>Duration of treatment</b> | 56 days |
| Study intervention | The screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. Part I is an open-label study, single center and dose escalation evaluation in six subjects. Six subjects will be initially evaluated for safety and efficacy assessments at low-dose (1 capsules TID) for 28 days. A safety checkpoint will be evaluated at day-28 for entering the high-dose (2 capsules TID). The subjects who pass the checkpoint will be initially evaluated for safety and efficacy assessments at high-dose (2 capsules TID) for 28 days. There will be an evaluation with all safety assessments data to decide whether this study passes the checkpoint to enter Part II. |




| Primary endpoint Secondary endpoints | <ul> <li>Improvement of 40% or greater in ADHD Rating Scale-Investigator Rated (ADHD-RS-IV) from baseline up to 8 weeks treatment</li> <li>Change from baseline in the Conners' Adult Attention- Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) to 8 weeks treatment.</li> <li>Clinical Global Impression-ADHD- Severity (CGI- ADHD-S) and Clinical Global Impression-ADHD- improvement (CGI-ADHD-I) score of 2 or lower.</li> </ul> |
|---|---|
| Safety Evaluation | A. Change from baseline in: 1. vital sign 2. physical examination 3. electrocardiogram (ECG) 4. laboratory tests (hematology and biochemistry) B. Incidence of AE/SAE C. Suicidal ideation and behavior by Columbia-Suicide Severity Rating Scale (C-SSRS) |
| Statistical method | Descriptive Statistics |




## LIST OF ABBREVIATIONS/DEFINITIONS

ADHD

Attention-Deficit/Hyperactivity Disorder

ADHD-RS-IV

Attention-Deficit/Hyperactivity Disorder Rating Scale-IV

AE

Adverse Events, whether or not considered related to the investigational drug, must be recorded in CRF.

CAARS-S:S

Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version

CGI-ADHD-I

Clinical Global Impression- Attention-Deficit/Hyperactivity Disorder –Improvement

CGI-ADHD-S

Clinical Global Impression- Attention-Deficit/Hyperactivity Disorder - Severity

CHO

Chinese Hamster Ovary

Clinical monitor

The designated CRA monitoring this study for the sponsor

CRA

Clinical Research Associate

CRC

Clinical Research Coordinator

CRF

Case Report Form

CRO

Contract Research Organization

C-SSRS

Columbia-Suicide Severity Rating Scale

• DSM-5

The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition

ECG

The Electrocardiogram (ECG) is a graphical recording of the cardiac cycle produced by an electrocardiograph.




HDL

**High-Density Lipoprotein** 

HPLC

High Performance Liquid Chromatography

ICF

Informed Consent Form

ICH-GCP

International Conference of Harmonization-Good Clinical Practice

• IEC

Independent Ethics Committee

IRB

Institutional Review Board

LDH

Lactate Dehydrogenase

• LDL

Lower-Density Lipoprotein

NET

Norepinephrine Transporter

• NLT

Not Less Than

NMT

Not More Than

NOAEL

No Observable Adverse Effect Level

• NRI

Norepinephrine Reuptake Inhibitor

PITDC

Medical and Pharmaceutical Industry Technology and Development Center

SAEs

Serious Adverse Event(s), whether or not considered as related to the investigational drug must be recorded and reported.

The serious adverse event is defined as following:

Death

Life-threatening condition

Inpatient hospitalization or prolongation of existing hospitalization




Persistent or significant disability/incapacity

Congenital anomaly/birth defect

Required intervention to prevent permanent impairment/damage

#### • Severity Rating of AE

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL†.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

†Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

#### • SHR

Spontaneous hypertensive rat

#### SOP

**Standard Operation Procedure** 

#### Study Cohort

The Study Cohort is defined as a group or cohort of subjects who are assigned to take the same dose level of the study drug.

#### • TID

Three times a day

#### WKY rat

Wistar-Kyoto rat

#### TLC

Thin Layer Chromatography




# 1. Background Information

### 1.1 Description of PDC-1421 Capsule

PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (*Polygala tenuifolia* Willd.) as active ingredient. Radix Polygalae is a traditional herb commonly prescribed in China to induce sedation, benefit the mentality and to promote expectoration. It has also been used for insomnia, anxiety, and heart palpitations<sup>1</sup>.

### 1.1.1 Preparation

Raw materials originated from *P. tenuifolia* were obtained from Shanxi, China. After having been cleaned and residual stems removed, the root was sun-dried and became the botanical raw material for producing the study drug (PDC-1421 capsule). Raw materials shall comply with physical/chemical specifications, and fingerprint determination via HPLC and TLC shall show desired contents. The materials shall comply with criteria for heavy metal, pesticide residues and aflatoxins to avoid contaminations. Acceptable raw materials were water extracted, partially purified by column chromatography, concentrated, and spray-dried to become the drug substance PDC-1421, a yellowish powder. The yield rate from raw materials to PDC-1421 is about 1.4%. Formulation and encapsulation of drug substance PDC-1421 produced the final product of PDC-1421 Capsule. Specifications of PDC-1421 Capsule are tabulated in Table 1.




Table 1. Specifications of PDC-1421 Capsule

| Test Items | Specifications |
|---|---|
| Physical | Vallavijsh Cramulas in brownish agnavla |
| Appearance | Yellowish Granules in brownish capsule. |
| Loss on Drying | NMT 6% |
| Water Extractives | NLT 80% |
| Dilute-Alcohol | NLT 70% |
| Extractives | INL1 7070 |
| Total Ash | NMT 5% |
| Acid-Insoluble Ash | NMT 4% |
| <b>Alcohol Extractives</b> | NLT 38% |
| | 1. One grayish blue band has same $R_f$ value as reference |
| TLC | standard (3',6-disinapoylsucrose); |
| | 2. One watchet blue band has same $R_f$ value as reference |
| | standard (Glomeratose A). |
| HPLC of markers | 1. $10.0 \text{ mg/g} \le \text{Glomeratose A} \le 30.0 \text{ mg/g}$ . |
| 2. $38 \text{ mg/g} \le 3',6\text{-Disinapoylsucrose} \le 95 \text{ mg/g}.$ | |
| UV Spectrum | $\lambda_{max}$ : 230 – 240 nm; 315 – 325 nm |
| IR Spectrum (cm <sup>-1</sup> , | Peak at: $3380 \pm 100$ Broad, $2938 \pm 20$ Sharp, $1605 \pm 10$ Sharp, |
| %T) | $1455 \pm 10 \text{ Sharp}, 833 \pm 10 \text{ Sharp}.$ |
| pH | Dissolved in distill deionized water at a concentration of 0.1 |
| pii | $g/ml$ , $3.8 \le pH \le 5.8$ . |
| Uniformity | 90-110% |
| Weight Variation | 90-110% |
| | Cu < 20 ppm, As < 1 ppm, |
| Heavy Metal | Pb < 5 ppm, Cd < 0.2 ppm, |
| | Hg < 0.1 ppm |
| | Total aerobic plate count: NMT 10 <sup>3</sup> CFU/g |
| | Mold and yeast count: NMT 100 CFU/g |
| Microbial Purity | Echerichia coli: Undetectable |
| | Staphylococcus aureus: Undetectable |
| | Salmonella: Undetectable |

NMT: not more than; NLT: not less than

PDC-1421 used in phase I clinical trial was manufactured at the Medical and Protocol




Pharmaceutical Industry Technology and Development Center (PITDC) in New Taipei City, Taiwan. In order to scale up the production and in compliant with GMP (Good Manufacturing Procedures), the producer has been changed to the Herbal Medicine GMP Plant of the Industrial Technology Research Institute (ITRI) in Hsinchu County, Taiwan. Products produced at ITRI Plant have been tested and meet defined specifications prior to use in this study.

### 1.1.2 Composition

Each PDC-1421 Capsule consists of 380 mg PDC-1421 drug substance and 20 mg of excipients. The composition of PDC-1421 Capsule is shown in Table 2.

Table 2. Composition of PDC-1421 Capsule

| Name of Ingredient | mg per Capsule | Function |
|--------------------|----------------|-------------------|
| PDC-1421 | 380 mg | Active ingredient |
| Silicon dioxide | 10 mg | Excipient |
| Magnesium stearate | 10 mg | Excipient |

### 1.1.3 Storage and Handling

During stability test, physical examination, loss on drying and contents assays of the characteristic markers (3',6-disinapoylsucrose and Glomeratose A) were conducted. The results indicated that PDC-1421 Capsule is stable when stored in a well-closed brown bottle at room temperature for at least 24 months.

# 1.2 Non-clinical Study of PDC-1421

Pharmacology studies were conducted at MDS Pharma Services, Taiwan. Nonclinical toxicity studies were conducted in accordance with Good Laboratory Practice at the Development Center for Biotechnology, Taiwan. Safety pharmacology studies were compliance with Good Laboratory Practice by Level Biotechnology, Inc. and Charles River Laboratory, Inc. Pharmacodynamics studies were conducted at PITDC, Taiwan.

### 1.2.1 Efficacy Pharmacology

Two *in vitro* studies and one *in vivo* study have been completed to evaluate pharmacological activities of PDC-1421.




#### 1.2.1.1 Radio-ligand Binding Assay

Radio-ligand binding assays were performed on 168 molecular targets, including receptors, ion channels and transporters, to discover the possible functional agonism and/or antagonism of PDC-1421 at concentration of 100  $\mu$ g/ml. Table 3 showed the result in this study, indicating that PDC-1421 specifically inhibited norepinephrine transporter. Other molecules, such as histamine receptor or cholinergic receptor, were not significantly influenced. The results suggested that PDC-1421 shall not induce side effects such as hypersomnia or dry month. Subsequent studies applying different concentration showed that the inhibition of norepinephrine transporter by PDC-1421 is dose-dependent, within 3 to 100  $\mu$ g/ml. Norepinephrine transporter inhibitors have been developed as the ADHD treatment, such as Atomoxetine. Therefore, PDC-1421 has the potential to be used as an ADHD medication. The subsequent studies were performed to investigate the activities of PDC-1421 used to treat ADHD.

Table 3. Summary of Significant Activities in radio-ligand binding assay

| Assay Name | IC <sub>50</sub> (μg/ml) |
|------------------------------------------|--------------------------|
| Norepinephrine Transporter (NET) Binding | 11.8 |

#### 1.2.1.2 Neurotransmitter Uptake Assay

Atomoxetine, which is one of ADHD medications on market, is a potent norepinephrine uptake inhibitor *in vitro* and *in vivo* with relatively low affinity for serotonin and dopamine uptake processes<sup>2,3</sup>. Uptake assays were conducted to study the effect of PDC-1421 on the reuptake of norepinephrine, serotonin and dopamine. The results of uptake assay are summarized in Table 4.


Table 4. Summary for neurotransmitter uptake assay

| Assay Name | Test Substance | Dose | Inhibition<br>% | IC <sub>50</sub> |
|---|---|---|---|---|
| Norepinephrine | PDC-1421 | $1 \mu g/mL$ | 52 | 0.70 μg/mL |
| Uptake | Desipramine | | | $0.44~\mu g/mL$ |
| — Орtаке<br>——— | | | | (1.66 nM) |
| Dopamine | PDC-1421 | $300~\mu g/mL$ | 55 | 246 μg/mL |
| Uptake | Nomifensine | | | $1.62~\mu g/mL$ |
| | | | | (6.83 nM) |
| Serotonin | PDC-1421 | 100 μg/mL | 52 | 107 μg/mL |
| Uptake | Fluoxetine | | | $0.87~\mu g/mL$ |
| _ | | | | (2.83 nM) |

PDC-1421 inhibited Norepinephrine reuptake at a 0.70  $\mu$ g/mL, much lower than of the concentration to inhibit dopamine (246  $\mu$ g/mL) or serotonin (107  $\mu$ g/mL). The results indicated that primary pharmacological effect of PDC-1421 may be with its norepinephrine reuptake inhibition, rather than serotonin or dopamine reuptake inhibition. The results are consistent with radio-ligand binding assay, indicated that PDC-1421 is highly specific in the inhibition of norepinephrine transporter.

#### 1.2.1.3 Tetrabenazine (TBZ)-induced Hypothermia Model

According to above assays, PDC-1421 is a selective norepinephrine reuptake inhibitor. A previous study has shown that the elevated concentration of norepinephrine produced by norepinephrine reuptake inhibitor (NRI) resulted in elevation of body temperature in reserpine-induced hypothermia animal model<sup>4</sup>. Reversed temperature in hypothermia model is an index to quantify the effect of NRI.

PDC-1421 was tested by the TBZ-induced hypothermia model to study the effect on norepinephrine reuptake inhibition. Vehicle, PDC-1421 and imipramine (positive control) were orally administrated to individual groups of experimental mice one hour before TBZ treatment, and body temperatures were recorded at appropriate time point. The results were summarized in Table 5.


Table 5. Summary for pharmacology study on norepinephrine reuptake inhibition.

| Tractment | Dose | % Inhibition in Body Temperature | | |
|---|---|---|---|---|
| Treatment | (mg/kg) | 60 min after TBZ | 90 min after TBZ | 120 min after TBZ |
| PDC-1421 | 10 | 5 | 0 | 0 |
| PDC-1421 | 30 | 30 | 33 | 27 |
| PDC-1421 | 100 | 55* | 59* | 63* |
| PDC-1421 | 300 | 77* | 74* | 80* |
| Imipramine | 3 | 89* | 84* | 83* |

<sup>\*</sup> The inhibition of TBZ-induced hypothermic response by  $\geq 50\%$  is considered as significant response

The results suggest that PDC-1421 at 100 mg/kg p.o. may be associated with NRI activity as evidenced by effect on TBZ-induced hypothermia in mice.

#### 1.2.1.4 Spontaneous hypertensive rat (SHR) Model

According to above assays, PDC-1421 is a selective norepinephrine reuptake inhibitor. Norepinephrine has also been proposed to play a key role in the pathophysiology and pharmacotherapy of ADHD<sup>5,6,7</sup>. The SHR is a valid and currently accepted model for the study of ADHD<sup>9</sup>. The SHRs are known to display hyperactivity, impulsivity, poor sustained attention, and deficits in learning and memory processes in comparison with normotensive Wistar-Kyoto (WKY) rats<sup>10</sup>. In order to proof of concept that PDC-1421 possesses the potential of treating ADHD, a local motor activity assay was performed by using SHR. Horizontal activity of SHR is recorded within one hour in Automated Locomotor Activity Analysis System Chamber. Intraperitoneal injection of 5 mg/kg atomoxetine, as a positive control, inhibited total activity of SHR rats significantly after 1 and 4 days administration. Atomoxetine is oral capsule in treatment usage. The course of treatment of atomoxetine needs one to three weeks for a good therapeutic response. The absorption of intraperitoneal injection is better than oral administration. PDC-1421 was designed as an oral drug substance. To determine PDC-1421's anti-ADHD effective dose, male SHR were orally given PDC-1421 dissolved in Saline at a dosage of 75, 225 or 675 mg/kg bodyweight at each exposure. The data revealed that oral administration of PDC-1421 for 1 and 4 days significantly inhibit total activity of SHR at the concentration of 675 mg/kg.




### Total Locomotor Activity



Figure 1. The local motor activity assay in different dose of PDC-1421.

Asterisk (\*) represents P-value <0.05 between control and treatment groups.

Double-asterisk (\*\*) represents P-value <0.01 between control and treatment groups.

### 1.2.2 Safety Pharmacology

In order to verify the possible adverse reactions, five studies were conducted to evaluate the effects of PDC-1421 on central nervous system, autonomic system, cardiovascular function, respiratory function, gastrointestinal system, renal function, allergy, inflammation, metabolism and hERG tail current assay:

- EfficacyProfiling in vivo®
- Safety Pharmacology Testing Package
- AdverseEventProfiling in vivo®
- Safety Pharmacology test in Central Nervous System, Cardiovascular System and Respiratory System
- hERG tail current assay

The significant findings were summarized in Table 6.




Table 6. Summary of the finding in safety pharmacology

| Study package | Study condition and findings |
|---|---|
| Efficacy Profiling | <ul> <li>Oral administration of PDC-1421 at 3000 mg/kg did not cause any significant change <i>in vivo</i> studies.</li> <li>PDC-1421 at 300 μg/ml did not demonstrate any significant activity (≥50% change) <i>in vitro</i> studies.</li> </ul> |
| Safety Pharmacology Testing Package | <ul> <li>PDC-1421 concentration at 300 μg/mL:</li> <li>Decrease in acetylcholine and BaCl<sub>2</sub>-induced constriction in guinea pig ileum.</li> </ul> |
| Adverse Event Profiling in vivo® | <ul> <li>PDC-1421 oral dose at 3000 mg/kg: <ul> <li>Inhibition of gastric emptying in fasted rats (-45%)</li> </ul> </li> <li>PDC-1421 oral dose at 3000 mg/kg for 7 days: <ul> <li>Increase in RBC on day 2 in blood chemistry</li> </ul> </li> <li>Increase in K<sup>+</sup> and decrease in glucose on day 2 in blood chemistry</li> <li>Decrease in LDH (lactate dehydrogenase) on day 8 in blood chemistry</li> </ul> |
| Safety Pharmacology<br>test in Cardiovascular<br>System | <ul> <li>RR interval elongation, heart rate decrease, diastolic arterial pressure decrease and increased sinoatrial arrest incidence were found in dogs in 2500 mg/kg group.</li> <li>Diastolic arterial pressure decrease was found in dogs in 2500 mg/kg group.</li> </ul> |
| hERG tail current assay | Below the dosage, 0.8 mg/ml PDC-1421, should be viewed as the "no effect concentration" in this assay. |

Few effects, including gastrointestinal effects, electrolytes equilibrium, blood sugar value, heart rate decrease and diastolic arterial pressure decrease were found in safety pharmacology. These findings provided scientific evidence in further clinical study to evaluate the influence of PDC-1421.


#### 1.2.3 Cytochrome P450 Interaction with PDC-1421

Cytochrome P450 (CYP450) enzyme assay was conducted for PDC-1421 to evaluate existence of potential drug interaction. The IC<sub>50</sub> values of each CYP450 isozymes are summarized in Table 7.

Table 7. Summary of IC<sub>50</sub> values of CYP450 isozymes

| CYP isozyme | Species | Concentration | Inhibition % | IC50 |
|-------------|---------|---------------|--------------|---------------|
| CYP 1A2 | Human | 100 μg/mL | 54 | $84 \mu g/mL$ |
| CYP 2C9 | Human | 100 μg/mL | 57 | $74 \mu g/mL$ |
| CYP 2C19 | Human | 100 μg/mL | 67 | 51 μg/mL |
| CYP 2D6 | Human | 100 μg/mL | 69 | 53 μg/mL |
| CYP 3A4 | Human | 100 μg/mL | 58 | 67 μg/mL |

A lower potential of causing drug-drug interaction was verified with lower CYP450 inhibition in this study.  $IC_{50}$  of CYP inhibition is higher than  $IC_{50}$  of *in vitro* pharmacological study (11.8 and 0.7 µg/mL in NET radioligand binding assay and reuptake assay, respectively), indicating that taking PDC-1421 with substrate of these CYP enzymes, including imipramine, paroxetine and warfarin, may not influence the blood concentration of these prescribed drugs.

### 1.2.4 Toxicology

Toxic effects of investigational drug are important considerations for human use. Several toxicology studies have been conducted to evaluate the toxic effects of PDC-1421.

### 1.2.4.1 Single Dose Acute Toxicity Study in Rats

Acute toxicity of test drug may predict effect of over dose. Four doses of PDC-1421 at 0, 1250, 2500 and 5000 mg/kg p.o. were given to different groups of rats. General demeanor, clinical signs, mortality, body weight and gross necropsy findings were evaluated and recorded. There has been no treatment-related pharmacological effect found with all 4 doses. Therefore, the "no observable adverse effect level" (NOAEL) is set at 5000 mg/kg in rats based on the results of this study.


#### 1.2.4.2 28-day Repeated Dose Subacute Toxicity Study in Rats

The duration of repeated dose toxicity study will be extrapolated to human therapeutic duration. Thus, toxic effects related to test drug dose in long term administration and determination of NOAEL are very important in further clinical study. Four groups of rats were administered with 0, 750, 1500 and 3000 mg/kg /once daily p.o. for 28 days respectively. Moribundity/mortality, clinical signs, body weight, food consumption, ophthalmology, clinical pathology (including urinalysis, hematology and serum chemistry), gross necropsy, organ weight and histopathology, were evaluated on those experimental rats. No death nor severe side effects had been observed. However, some effects were considered treatment-related as shown in Table 8:

Table 8. Summary of 28-day repeated dose toxicity study in rats

| Group | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| Dose (mg/kg/day) | 0 | 750 | 1500 | 3000 |
| Male | | | | |
| Calcium (mg/dL) <sup>1</sup> | $10.7\pm0.7$ | $10.8 \pm 0.8$ | $10.4 \pm 0.9$ | $9.6 \pm 0.5^*$ |
| Female | | | | |
| Sodium (mEq/L) <sup>2</sup> | $147.4 \pm 1.8$ | $148.1 \pm 1.6$ | $147.8 \pm 1.8$ | $150.5 \pm 2.1^*$ |
| Thymus weight (mg) | $501.3 \pm 122.9$ | $449.4 \pm 91.7$ | $418.4 \pm 66.7$ | $377.2 \pm 81.2^*$ |

Reference range: 1: 10.5~12.2; 2: 136~156

Concluded by the investigating institute, those abnormal are mild and did not influence the physical condition of experimented rats. Therefore, NOAEL for PDC-1421 in rats under this study condition is 3000 mg/kg/day.

#### 1.2.4.3 28-day Repeated Dose Subacute Toxicity Study in Dogs

In order to determine NOAEL in dogs, PDC-1421 was repeatedly administered to four groups of dogs at dose levels of 0, 300, 1000, 3000 mg/kg once daily for 28 days. Soft feces were found in male dogs at 3000 mg/kg. There are several differences of physical value, lower mean corpuscular volume and monocytes in males and lower cholesterol and triglyceride in females, between test groups and control group, but these effects are not treatment-related or dose-dependent and within DCB (Development Center for Biotechnology) historical data range. Therefore, NOAEL for PDC-1421 in dogs is set at 3000 mg/kg.

<sup>\*:</sup> *p* < 0.05




#### 1.2.4.4 Genotoxicity

Three studies, including Ames test, micronucleus test and chromosome aberration assay, were conducted to evaluate the genotoxicity of PDC-1421. In Ames test, five different strains of *Salmonella typhimurium* were used to evaluate the mutagenic potential when incubated at different concentration of PDC-1421. No mutation induced by PDC-1421 was observed. In micronucleus test, three doses of PDC-1421 at 500, 1000, 2000 mg/kg p.o. were administered to three different groups of BALB/c mice and the ability of PDC-1421 to induce micronucleated reticulocytes in mouse peripheral blood was measured. The results of this study indicated that PDC-1421 posed-negative response to clastogenic micronucleated reticulocytes in mice. In chromosome aberration assay, clastogenic activity was evaluated in Chinese hamster ovary (CHO) cells after adding the different concentration of PDC-1421. Based on the results of this study, chromosomes in CHO cells are not affected by PDC-1421. In conclusion, PDC-1421 does not pose any risk of genotoxicity.

### 1.3 Results of Phase I Clinical Trial Study of PDC-1421

In phase I trial, all total of 85 subjects were screened at study site and 30 subjects were enrolled. They were 9 subjects in cohort A with 7 administered PDC-1421 (380 mg) and 2 administered placebo, 1 of 7 PDC-1421 subjects (P01) had no laboratory test data at baseline; 8 subjects in cohort B with 6 administered PDC-1421 (1140 mg) and 2 administered placebo; 4 subjects in cohort C with 3 administered PDC-1421 (2280 mg) and 1 administered placebo; 9 subjects in cohort D with 7 administered PDC-1421(3800 mg) and 2 administered placebo, 1 of 7 PDC-1421 subjects (P27) had abnormal laboratory data at screening visit.

Physical examination was determined to be "normal" on every Body System in each cohort and no subject had DLT and toxicity grade.

All of the changes of vital signs from baseline of PDC-1421 and placebo group were mild and did not exceed the limit of normal range. Furthermore, all of the toxicity grades of vital signs were the lowest, systolic blood pressure in grade 1, increase >20 mm/Hg than baseline at 4 hours. No medical intervention/therapy was required. There was no correlation of changes from baseline or changes in the toxicity grade of vital signs between doses of PDC-1421.

All changes of laboratory test data from baseline of PDC-1421 group were mild and no clinically significant deviation from the normal range. Furthermore, the toxicity grades




of laboratory test data of PDC-1421 and placebo groups were the lowest, grade 1. No medical intervention/therapy was required. There was no correlation of change from baseline or change in the toxicity grade of laboratory test between doses of PDC-1421. Only two grade 2 toxicity (at 24 hours in glucose in cohort A and at 4 hours in glucose in cohort B) occurred in placebo group and no medical intervention/therapy were required for these cases.

ECG was determined to be "normal" in each time point and in each cohort. No subject had DLT and toxicity grade.

C-SSRS were all 0 point on Suicidal ideation, Intensity of ideation, Suicidal behavior in each cohort.

No subject had serious adverse event and no subject discontinued due to adverse event, no clinically significant finding in physical examinations, vital signs, electrocardiogram, laboratory measurements, and C-SSRS was observed throughout the treatment period, and the oral administration of PDC-1421 in healthy volunteers was safe and well-tolerated for the dose from 380 mg to 3800 mg. During the treatment period, five subjects reported to experience eight mild adverse events shown as Table 9. The severity of these eight adverse events was all mild and no medical action required. There was no correlation between number, severity, relationship and outcome of adverse events found between doses of PDC-1421 and placebo. Further, there was no clinically significant finding in electrolyte level and gastrointestinal discomfort during monitoring in the clinical trial. There were two mild adverse events such as lower heart rate and higher systolic blood pressure. In the dog telemetry study, only lower heart rate was found but not higher systolic blood pressure.

Table 9. Frequencies of Adverse Events

| Adverse events | Frequency | | | | |
|---|---|---|---|---|---|
| BODY System | Cohort A | Cohort B | Cohort C | Cohort D | Placebo |
| | (380 mg) | (1140 mg) | (2280 mg) | (3800 mg) | N=7 |
| | N=7 | N=6 | N=3 | N=7 | |
| Digest System | 3/7 | 0 | 0 | 0 | 1/7 |
| FLATULENCE | 2/7 | 0 | 0 | 0 | 1/7 |
| CONSTIPATION | 1/7 | 0 | 0 | 0 | 0 |
| Nervous System | 0 | 0 | 2/3 | 0 | 2/7 |
| SOMNOLENCE | 0 | 0 | 1/3 | 0 | 2/7 |
| STOMATITIS<br>ULCER | 0 | 0 | 1/3 | 0 | 0 |




### 1.4 Potential Risk and Benefit

#### 1.4.1 Potential Risk

The toxicological profile of PDC-1421 was characterized in single and repeat oral dose studies of up to 28 days in rats and repeat oral dose studies of up to 28 days in dogs. Genetic toxicology and safety pharmacology have also been conducted. PDC-1421 was observed to be associated with some adverse effects in serum electrolytes and GI function, but none were clinically significant. Therefore, potential risks of PDC-1421 are fluctuated electrolyte level and gastrointestinal discomfort. We monitored these in the Phase I study and there was no deviation of electrolyte level and no significant gastrointestinal discomfort during monitoring in the clinical trial. However, there were non-clinically significant mild lower diastolic blood pressure and lower heart rate in dog telemetry study and it has been only with the 2500 mg/kg, which is around the NOAEL for dogs. The cardiovascular systems will be monitored in the clinical study.

#### 1.4.2 Potential Benefit

According to nonclinical study results, the results of two *in vitro* assays support the fact that PDC-1421 is a selective norepinephrine reuptake inhibitor and have low affinity to serotonin and dopamine. A SHR animal model has shown that PDC-1421 has potential to develop as an ADHD medication. Furthermore, PDC-1421 will not pose the adverse effects caused by the molecules which possess anticholinergic or antihistamine activities due to its selectivity on norepinephrine transporter.

#### 1.4.3 Risk Benefit Ratio

Potential risks in nonclinical results outlined above are minor and easy to monitor. As there were adverse events in phase I trial, no similar findings were found in nonclinical studies. The subsequent trial could be benefited from gathering further safety information for PDC-1421 treatment.

# 1.5 Dosage Regimen

Based on the FDA's guidance documents, NOAELs from toxicity studies were used to estimate the starting dose in our study. Table 10 summarizes the MRSD for 60 kg human/day calculated from the NOAEL of 28 day repeating dose studies in rats and in dogs using safety margin at 75-fold.


Table 10. Calculation of starting dose

| Study | Species | Dosage | HED | Dose for 60 kg<br>human/day |
|---|---|---|---|---|
| 28-day repeated dose subacute oral toxicity study in rats | rat | 3000 mg/kg<br>(NOAEL) | 483.9 mg/kg | 387 mg/day<br>(MRSD) |
| 28-day repeated dose subacute oral toxicity study in dogs | dog | 3000 mg/kg<br>(NOAEL) | 1666.7 mg/kg | 1333 mg/day<br>(MRSD) |

Based on these calculations, we proposed the starting dose of PDC-1421 to be at 380 mg/day. In the phase I study, a single dose of PDC-1421 (oral administration) was used to evaluate the safety when taken by healthy subjects. The starting dose and dosage regimen are:

380 mg PDC-1421 (one capsule of PDC-1421 Capsule) once daily after meal

The dose escalation is as follows.

Cohort A (one capsule; 380 mg):

Cohort A enrolled nine subjects. Seven subjects received PDC-1421 Capsule and two received placebo. There was only one of placebo subjects who met a DLT due to the glucose value at 24 hours after drug administration. We continued the study to the next higher dosage, cohort B.

Cohort B (three capsules; 1140 mg):

Cohort B enrolled eight subjects. Six subjects received PDC-1421 Capsule and two received placebo. There was only one of placebo subjects who met a DLT due to the glucose value at 4 hours after drug administration. We continued the study to the next higher dosage, cohort C.

Cohort C (six capsules; 2280 mg):

Cohort C enrolled four subjects. Three subjects received PDC-1421 Capsule and one received placebo. There was no DLT in this cohort. We continued the study to the next higher dosage, cohort D.

Cohort D (ten capsules; 3800 mg):

Cohort D enrolled nine subjects. Seven received PDC-1421 Capsule and two received placebo. There is no DLT in the final cohort.

Based on the results, the maximum tolerated dose (MTD) is  $\geq 3800$  mg of PDC-1421 Capsule so that the safe and well-tolerated for PDC1-421 Capsule is from 380 mg to 3800 mg.

Protocol




According to studies in mouse model system to evaluate efficacious dose, SHR animal model, PDC-1421 was indicated to be efficient at oral administration of 675 mg/kg doses which are equivalent to about intraperitoneal injection of 5 mg/kg atomoxetine. The consideration is the course of treatment of atomoxetine, ADHD medication which is also a selective NRI, need one to three weeks for a good therapeutic response. There will be lower effective dose with long-term administration. The positive control, atomoxetine administrated by intraperitoneal injection in SHR animal model, and the absorption is better than oral. Base on the bioavailability is 63%, and the minimum starting dose is 0.5 mg/kg of Strattera (the trade name of atomoxetine), we translate the starting dose of PDC-1421 is 42.56 mg/kg (675 [mg] \* 63% \* 0.5 [mg/kg] / 5 [mg/kg] = 42.56 mg) and the human equivalent dose is about 2553.59 mg in 60 kg weight.



According to the result of phase I trial and preclinical study with SHR animal model, we choose 1140 mg (3 capsules) and 2280 mg (6 capsules) as the dosage regimen of Phase II trial.

# 1.6 Compliance with Protocol, Good Clinical Practice (GCP)

# and Applicable Requirement

This study and all operating procedures will be conducted in accordance with GCP guidelines, protocol and all applicable regulatory requirements issued by US FDA, to protect the rights, safety and well-being of the studying subjects.

# 1.7 Description of the Population to be Studied

We chose patients with Attention Deficit Hyperactivity Disorder as our subjects in this phase II trial.




# 2. Trial Objective

The primary objective of this trial was to determine the effective doses and treatment period of PDC-1421 Capsule in subjects with ADHD. The secondary objective was to evaluate the safety of PDC-1421 Capsule in subjects receiving PDC-1421at various dose levels.

# 3. Trial Design

## 3.1 General Design

Table 11. Summary of general design

| | Doub I |
|--------------|--------------------------------------------------|
| | Part I |
| Design | Open label, single center, dose escalation study |
| ADHD | 6 |
| patients | |
| Treatment | (1) Low dose: 1 capsule TID, 28 days |
| | (2) Checkpoint #1 |
| | (3) High dose: 2 capsules TID, 28 days |
| | (4) Checkpoint #2 |
| Assessment | Low dose: Once a week |
| interval | High dose: Biweekly |
| Efficacy and | Safety evaluation |
| safety | Efficacy evaluation |
| evaluation | |

The Screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The targeted population of this Part I study is six subjects who met the intent-to-treat basis.

Part I study is an open-label study, single center and dose escalation evaluation in six patients.

<u>Low dose</u>: Six subjects will be initially evaluated for safety and efficacy assessments at low-dose (1 capsule TID) for 28 days. Subject will return for visit once a week during treatment period.

Protocol




<u>Checkpoint #1</u>: There will be an evaluation with all safety assessments data to decide whether you pass the checkpoint to enter high-dose treatment or continue to receive a low-dose treatment by the investigator.

High dose: The subjects who pass the checkpoint #1 will be initially evaluated for safety and efficacy assessments at high-dose (2 capsules TID) for 28 days. Subject will return for visit biweekly during treatment period.

<u>Checkpoint #2</u>: There will be an evaluation with all safety assessments data to decide whether this study passes the checkpoint to enter Part II by the investigators.

Figure 2. General design of procedure Part I. Study.






## 3.2 Primary Endpoint

Improvement of 40% or greater in ADHD Rating Scale-Investigator Rated (ADHD-RS-IV) from baseline up to 8 weeks treatment.

# 3.3 Secondary Endpoint

Table 12 The secondary efficacy endpoints

| Number | Items |
|---|---|
| 1 | Change from baseline in the Conners' Adult Attention- |
| | Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version |
| | (CAARS-S:S) up to 8 weeks treatment. |
| 2 | Clinical Global Impression-ADHD- Severity (CGI-ADHD-S) and |
| | Clinical Global Impression-ADHD- improvement (CGI-ADHD-I) score |
| | of 2 or lower. |

# 3.4 Randomization and Blinding

Table 13. Summary of randomization and blinding

| | Part I |
|---------------|-------------------|
| Randomization | None (open label) |
| Blinding | None (open label) |

# 3.5 Investigational Drug

Investigational drug (PDC-1421 Capsule) will be maintained and dispensed by UCSF Medical Center. No one but the Investigator and/or his/her designee is permitted to access the investigational drug.

### 3.5.1 Dosage Form and Strength

PDC-1421 Capsule: 380 mg PDC-1421/capsule

#### 3.5.2 Manufacturer

ITRI (Industrial Technology Research Institute), Hsinchu County, Taiwan

#### 3.5.3 Route of Administration

Oral administration




### 3.5.4 Dosing Regimen, packing and labeling

### 3.5.4.1 Dosing Regimen

#### **Part I Study:**

Subjects will receive a low-dose treatment with 1 PDC-1421 Capsule thrice daily for 28 days (4 weeks). After passing a dose-up checkpoint for the safety of individual subjects, they will receive a high-dose treatment with 2 PDC-1421 Capsules thrice daily for another 28 days (4 weeks).

Dosing regimen for the study is summarized with drug packing on Table 14.

#### 3.5.4.2 Packaging

Investigational drug (PDC-1421 Capsule) are provided by BioLite, Inc. and stored in the UCSF Medical Center. Subjects will receive the investigational drug at each visit and also be requested to return unused drug at each visit. Drug packing for each part of the study is summarized with dosing regimen on Table 14.

#### **Part I Study:**

- Low-Dose: Subjects will receive a drug bag with 21 PDC-1421 Capsules each visit. A total 5 weekly visits will be requested during this 28-day treatment period.
- ➤ **High-Dose:** Subjects will receive 1 drug bag of 84 PDC-1421 Capsules/bag each visit. A total 3 biweekly visits will be requested during this 28-day treatment period.

Table 14. Summary of dosing regimen and packaging

| Part no. | | Part I | |
|---|---|---|---|
| Dosing/Ar | m | Low-Dose High-Dose | |
| Treatment | Duration | 28 days + 28 days | |
| Dosing | Placebo | N/A | N/A |
| Regimen | PDC-1421 | 1 Cap. TID | 2 Caps. TID |
| Packaging | | 21 PDC-1421 Caps./bag 84 PDC-1421 Caps./bag | |
| Visit Frequ | uency | Weekly Biweekly | |
| No. of Drug bags<br>Received / Visit | | 1 | 1 |
| Received / | Visit | | |




#### **3.5.4.3** Labeling

The drug bag of investigational drug will be clearly labeled as following:

For Part I-low dose (380 mg TID):

Test Drug: PDC-1421 Capsule

Amount: capsules ( reserved capsules included)

Subject Number: Drug Pack Number:

Study Protocol: BLI-1008-001 Drug Appearance: Brown capsule

Major Component: Each capsule contains 380 mg of PDC-1421

Dosing: 1 capsule thrice daily after meal for OO days and with extra OO days for reserved

Storage Condition: Store at a dry place at room temperature  $(15\sim25^{\circ}\text{C})$ 

Lot Number:

Manufacturer: Industrial Technology Research Institute

Date of Manufacture: Date of Expiration: Sponsor: BioLite, Inc.

Clinical Site: UCSF Medical Center

"Caution: New drug - Limited by Federal Law to investigational use".

注意:試驗新藥僅限特定臨床試驗使用

試驗藥物: PDC-1421 膠囊

數量: 顆膠囊 (含 顆備用膠囊)

藥物編號: 受試者編號: 回診次別: Visit

計劃書編號: BLI-1008-001

藥物外觀: 棕色膠囊

主成份: 每顆膠囊含有 380 mg PDC-1421

劑量:三餐飯後服用1顆膠囊,OO 日份 (外加 OO 日備用藥)

儲存條件: 儲存於乾燥常溫之環境 (15~25℃)

批號:

製造商: 工業技術研究院

製造日期: 有效日期:

廠商: 萊特先進生醫股份有限公司

試驗機構: 加州大學舊金山分校醫學中心

"Caution: New drug - Limited by Federal Law to investigational use".

注意:試驗新藥僅限特定臨床試驗使用




#### For Part I-High dose (760 mg TID):

Test Drug: PDC-1421 Capsule

Amount: capsules ( reserved capsules included)

Subject Number: Drug Pack Number:

Study Protocol: BLI-1008-001 Drug Appearance: Brown capsule

Major Component: Each capsule contains 380 mg of PDC-1421

Dosing: 2 capsules thrice daily after meal for OO days and with extra OO days for reserved

Storage Condition: Store at a dry place at room temperature (15~25°C)

Lot Number:

Manufacturer: Industrial Technology Research Institute

Date of Manufacture: Date of Expiration: Sponsor: BioLite, Inc.

Clinical Site: UCSF Medical Center

"Caution: New drug - Limited by Federal Law to investigational use".

注意:試驗新藥僅限特定臨床試驗使用

試驗藥物: PDC-1421 膠囊

數量: 顆膠囊 (含 顆備用膠囊)

藥物編號: 受試者編號: 回診次別: Visit

計劃書編號: BLI-1008-001

藥物外觀: 棕色膠囊

主成份: 每顆膠囊含有 380 mg PDC-1421

劑量: 三餐飯後服用 2 顆膠囊, OO 日份 (外加 OO 日備用藥)

儲存條件: 儲存於乾燥常溫之環境 (15~25℃)

批號:

製造商: 工業技術研究院

製造日期: 有效日期:

廠商: 萊特先進生醫股份有限公司

試驗機構: 加州大學舊金山分校醫學中心

"Caution: New drug - Limited by Federal Law to investigational use".

注意:試驗新藥僅限特定臨床試驗使用




### 3.5.5 Study Drug Storage

Investigational drugs will be stored in a locked cabinet at room temperature (15~25°C) in Department of Pharmacy, UCSF Medical Center.

# 3.6 Premature Termination or Suspension of the Study

The Investigator and/or the Sponsor may decide to stop the trial if:

- Safety assessment clearly indicates that one study arm is associated with more severe or serious adverse experiences.
- The Sponsor decides to terminate the trial if necessary.




# 4. Subjects Selection and Withdrawal

Inclusion and exclusion criteria in part I are as follows.

#### 4.1 Inclusion Criteria

- 1. Aged 18-70 years
- 2. Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study
- 3. Subjects must be able to understand and willing to sign informed consent
- 4. Able to discontinue the use of any psychotropic medications for the treatment of ADHD symptoms at screening
- 5. Meet strict operational criteria for adult ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
- 6. A total score of 20 or higher on the 12-item ADHD index of Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) at screening
- 7. Have a moderate or severe symptom of ADHD with score of 4 or higher in Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) at screening

### 4.2 Exclusion Criteria

- 1. Have any clinically significant concurrent medical condition (endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, anorexia, obesity or malignancy) that has become unstable and may interfere with the interpretation of safety and efficacy evaluations
- 2. Have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at screening that, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations
- 3. Have known serological evidence of human immunodeficiency virus (HIV) antibody
- 4. Are pregnant as confirmed by a positive pregnancy test at screening
- 5. Have QTc values >450 msec at screening using Fridericia's QTc formula
- 6. Have current of bipolar and psychotic disorders




7. Have a current major depression disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder and eating disorder (also if treated but not currently symptomatic)

**NOTE:** Comorbid diagnoses identified during screening and baseline are acceptable provided that ADHD is the primary diagnosis and the comorbid diagnoses will not confound study data or impair subject's ability to participate (per the Investigator's judgement and documented in source note).

- 8. Have any history of a significant suicide attempt, or possess a current risk of attempting suicide, in the investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS).
- 9. Have a history of jailing or imprisonment in the past 6 months due to worsening of symptoms of ADHD.

# 4.3 Subject Recruitment and Screening

At Visit 1, Investigator will introduce the proposed clinical study to subjects who are interesting in this study. If a subject is willing to undergo an informed consent process based on GCP and participate in this study, the subject will be examined as described in section 5.2. At Visit 2, based on Visit 1 measurements, subject who meets the recruitment criteria will be enrolled in this study.

# 4.4 Subject Identification

In order to protect each subject's privacy, only subjects' initials will be used as part of subjects' identifications. In addition, a subject number will be assigned to each subject who signed the ICF and each subject who is eligible to enroll in the study.



#### 4.4.1 Subject Initial Allocation

A subject's initial will be assigned to each subject by the clinical research coordinator (CRC). Remain blank in the 3<sup>rd</sup> and 4<sup>th</sup> space if there have no more initial(s) to be filled in.



#### 4.4.2 Subject Number Allocation

Each subject will be assigned a number by the CRC. All subject numbers will have eight digits.



The first digit: the part number; Part I will be assigned to "1", Part II will be assigned to "2".




## 4.5 Early Withdrawal of Subjects

Subjects will be withdrawn from this trial if they meet one of the following withdrawal criteria:

- Subjects wish to withdraw. (Subjects are not obligated to give reasons for discontinuation from this trial.)
- Subjects can't obey the regulation of the study.
- Investigator considers that withdrawal from study is the best interest of a subject.
- The subject is pregnant during the trial.

Subjects withdrawn from the study due to adverse event(s) must be followed until the events are recovered, recovered with residual effects, death, or lost to follow-up.

# 5. Treatment of Subjects

## 5.1 Description of Study Drug

PDC-1421 Capsule is a botanical investigational new drug. Each PDC-1421 Capsule contains 380 mg PDC-1421 drug substance extracted from dry root of *P. tenuifolia*. The detailed information of PDC-1421 Capsule is described in section 1.1.

#### 5.2 Treatment Schedule

Potential subjects will be introduced by Investigator of the study design at Screening. If the subject agrees to participate and signs the consent form, the screening process will begin. Suitability of the subject will be evaluated by inclusion/exclusion criteria.

In part I Study, six eligible subjects will receive a low-dose treatment with 1 PDC-1421 Capsule thrice daily for 28 days (4 weeks) and be assessed once a week (Visit 2, 3, 4, 5, and 6). After passing a dose-up checkpoint for the safety of individual subjects, these subjects will then receive a high-dose treatment with 2 PDC-1421 Capsules thrice daily for another 28 days (4 weeks). Subjects will be assessed every two weeks (Visit 6, 7 and 8) in high-dose treatment. After the end of part I Study, subjects will be requested to return for a follow-up visit (Visit 9) two weeks later after the last dose.

During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be




documented.

Table 15. Part I-schedule of assessments

| Procedure table: BLI-1008-001 protocol | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| *Week | -2 | 0 | 1 | 2 | 3 | 4 | 6 | 8 | 10 |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| DSM-V | $\checkmark$ | | | | | | | | |
| CAARS-S:S | $\checkmark$ | | | $\sqrt{}$ | | $\sqrt{}$ | $\sqrt{}$ | | |
| CGI-ADHD-S | $\checkmark$ | | | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | | |
| CGI-ADHD-I | | | V | V | V | V | | V | |
| ADHD-RS-IV | $\checkmark$ | | | $\sqrt{}$ | | $\sqrt{}$ | $\sqrt{}$ | | |
| C-SSRS | $\sqrt{}$ | | √ | $\sqrt{}$ | V | $\sqrt{}$ | | | |
| AE/SAE evaluation | | | √ | √ | √ | √ | √ | √ | |
| Concomitant | $\checkmark$ | | | $\sqrt{}$ | | $\sqrt{}$ | | | |
| Medication | | | | | | | | | |
| Physical | $\sqrt{}$ | | | | | | | | |
| examination | | | | | | | | | |
| Vital sign | $\sqrt{}$ | $\sqrt{}$ | | $\sqrt{}$ | | $\sqrt{}$ | $\sqrt{}$ | | |
| ECG | $\sqrt{}$ | | | | | | | | |
| Hematology | $\sqrt{}$ | $\sqrt{}$ | | $\sqrt{}$ | | $\sqrt{}$ | $\sqrt{}$ | $\sqrt{}$ | |
| <b>Blood Chemistry</b> | $\sqrt{}$ | | | √ | | √ | $\sqrt{}$ | | |
| Blood drawing | $\sqrt{}$ | | | √ | | √ | | √ | |
| (venipuncture) | | | | | | | | | |
| Pregnancy test | $\sqrt{}$ | | | | | | | | |

<sup>\*</sup>On  $\pm 2$  days.

## **5.2.1 Screening Phase (Visit 1)**

The Screening phase will be done within 1-2 weeks period and intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The items of physical, rating scales and laboratory examination at screening are outlined below:

- Informed consent
- Subject information, including date of birth, gender, body height and weight
- Medical history (within six month), including any clinically significant psychiatric, neurological, gastrointestinal, renal, hepatic, cardiovascular, respiratory, metabolic,




endocrine, hematological or other major disorders

- Pregnancy test
- Physical examination: skin, head, neck, eyes, ears, nose, throat, heart, lungs, abdomen (liver, spleen), neurological examination, lymph node and extremities.
- Vital sign: heart rate, blood pressure, body temperature
- ECG
- Hematology: RBC, WBC, platelets, hematocrit, hemoglobin, prothrombin time (PT), partial thromboplastin time (aPTT)
- Blood chemistry: AST, ALT, LDH, total bilirubin, BUN, serum creatinine, free thyroxine (FT4), TSH, sodium, calcium, potassium, HbA1c, LDL, HDL, triglyceride, cholesterol
- DSM-5, CAARS-S:S, CGI-ADHD-S, ADHD-RS-IV, C-SSRS
- Concomitant medication evaluation
- Eligibility evaluation: laboratory data, other tests and evaluation results shall be obtained at Screening to determine the appropriateness of subject enrolled in this study

# 5.2.2. Part I Study. - Treatment Period (Visit 2~8) and Follow-up (Visit 9)

Subjects who meet the eligibility criteria will be enrolled and take test drug at this period. Six eligible subjects will take 1 capsule of PDC-1421 Capsule thrice daily for four weeks. They will receive a drug bag and be instructed to take 1 PDC-1421 Capsule thrice daily after meals. Weekly visits (Visit 2, 3, 4 and 5) will be requested during this 28-day treatment period. At Visit 6, all subjects will be evaluated with safety assessments and to be decided whether they will enter the high-dose treatment by the investigator. In the high-dose treatment, subjects will receive a drug bag and be instructed to take 2 PDC-1421 Capsule thrice daily after meals for 4 weeks. Biweekly visits (Visit 6, 7 and 8) will be requested during this 28-day treatment period. After two weeks of the last dose administration, subjects are assessed for a follow-up. Then, a checkpoint will be conducted. If subjects have no drug-related SAE, the schedule can be conducted to the part II. The items of safety and efficacy parameters at treatment period are outlined below:

- Physical examination: skin, head, neck, eyes, ears, nose, throat, heart, lungs, abdomen (liver, spleen), neurological examination, lymph node and extremities (only at Visit 8).
- Vital sign: heart rate, blood pressure, body temperature




- ECG (Only at Visit 8).
- Hematology: RBC, WBC, platelets, hematocrit, hemoglobin, prothrombin time (PT), partial thromboplastin time (aPTT) (Only at Visit 2,4,6,7 and 8).
- Blood chemistry: AST, ALT, LDH, total bilirubin, BUN, serum creatinine, free thyroxine (FT4), TSH, sodium, calcium, potassium, LDL, HDL, triglyceride, cholesterol (Only at Visit 2,4,6,7, and 8).
- CAARS-S:S, CGI-ADHD-S, CGI-ADHD-I, ADHD-RS-IV, C-SSRS and concomitant medication evaluation.
- AE/SAE evaluation (Subjects will not need to be assessed for AE/SAE at visit 2.)
- Drug accountability

Follow-up visit will be performed at visit 9 after two weeks of the last dose administration. The test items are outlined in the following:

- C-SSRS.
- AE/SAE evaluation
- Pregnancy test

#### 5.3 Other Medication During the Study

To avoid conflict or unknown effects with the study drug, subjects are prohibited from taking any anti-ADHD medication and psychoactive drugs, as per the exclusion criteria, including MAOIs (monoamine oxidase inhibitor), NRIs (norepinephrine reuptake inhibitor) and norepinephrine receptor agonist/antagonist. Subjects can't combine the newly-initiated psychotherapy. If subjects have severe insomnia and are currently taking Zolpidem, Zopiclone or Zaleplon (sedative-hypnotics), they will be queried whether they can comply with the discontinuation:

- 1. Subjects who indicate that they can discontinue will be washed out for 1 week, and then allowed to begin study protocol;
- 2. Subjects who indicate that they are unable to discontinue will be allowed to enroll if they are able to agree that their use will be consistent and will not change for the duration of the study. (The maximum daily dose in Zolpidem, Zopiclone and Zaleplon are 10 mg, 7.5 mg and 10 mg respectively.)




# 6. Efficacy Assessments

# 6.1 Specification of the efficacy parameters

Efficacy parameters are outlined as follows:

- ADHD-RS-IV
- Clinical Global Impression
- CAARS-S:S

## 6.2 Methods and Timing for Assessing, Recording, and

#### Analyzing of Efficacy Parameters.

The data obtained from eligible subjects before study drug administration in Visit 2 are set as baseline. After the beginning of treatment, the collection of data of efficacy parameters are performed at planned treatment schedule as section 5.2. CRC shall record these data in CRF in detail after each visit during the treatment period. In part I study, efficacy assessments are conducted from screening stage to the last visit. The rating scales are as follows:

#### ADHD-RS-IV

The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR' criteria for ADHD that provides a rating of the severity of symptoms<sup>15</sup>. The adult prompts serve a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible total score of 0–54. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often. Clinicians should score the highest score that is generated for the prompts for each item

For inattention (IA) subscale raw score: Add the odd-numbered 9 items

For hyperactivity-impulsivity (HI) subscale raw score: Add the even-numbered 9 items

To obtain the total raw score: Add the IA and HI subscale raw scores.




#### • Clinical Global Impression

At the baseline visit, clinicians completed the CGI-S and were asked to evaluate the severity of subjects' illness with respect to ADHD symptoms based on the clinician's experience with this particular population. Possible scores ranged from 1 (normal, not ill at all) to 7 (among the most extremely ill subjects). At all subsequent study visits, clinicians used the CGI-I to rate the subjects' total improvement based on comparison with their baseline assessment from 1 (very much improved) to 7 (very much worse).

#### CAARS-S:S

Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (Conners et al., 1998; CAARS-S:S). This consists of 26 items rated from 0 'not at all, never' to 3 'very much, very frequently.' Four subscales each composed of 5 items (A: inattention/memory problems; B: hyperactivity/restlessness; C: impulsivity/emotional lability; and D: problems with self-concept) as well as a 12-item ADHD index can be computed<sup>14</sup>. The CAARS-S:S was administered by computer-assisted personal interview (CAPI) prior to the first treatment session.




# 7. Safety Assessments

## 7.1 Specification of Safety Parameters

Safety parameters are outlined as follows:

- Data collected from the physical examinations, vital sign, ECG and laboratory test in scheduled visit
- Adverse events reported
- Serious adverse events reported
- C-SSRS evaluation

## 7.2 Methods and Timing for Assessing, Recording, and

## **Analyzing of Safety Parameters**

The data obtained before study drug administration in Visit 2 are set as baseline. After the beginning of treatment, the collection of data of safety parameters are performed at planned treatment schedule as section 5.2. AE or SAE will be closely monitored during the study period. CRC shall record these data in CRF in detail. In part I, data are recorded from screening stage to the last visit.

## 7.3 Adverse Events (AEs)

Adverse event is any unfavorable and unintended symptom, syndrome, medical condition or experience that develops or worsens within the study period. In this Phase II trial, any clinically significant abnormal findings, including causing the subject to withdraw from the study, requiring treatment or causing apparent clinical manifestations, or judged relevant by the investigator, are considered to be AEs and will be monitored and recorded. AE may not be causal relationship with study medication or clinical study. Whether related to study medication or not, CRC shall record the information of AEs in CRF. The information of AEs contains characteristic, onset and duration, frequency, the Investigator's opinion of the relationship to the study drug (unrelated, unlikely, possibly, probably, definitely), outcome (recovered, recovered with residual effects, continuing, death, lost to follow-up) and severity. Common Terminology Criteria for Adverse Events v4.03 (CTCAE Table 16) is a descriptive terminology and the grading (severity) scale is provided for each AE term.


Table 16. Common Terminology Criteria for Adverse Events

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL†. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE.‡ |

<sup>\*</sup>Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

#### 7.4 Serious Adverse Events (SAE)

SAE is defined as any significantly untoward medical occurrence, including:

- Death
- Life-threatening condition
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect
- Required intervention to prevent permanent impairment/damage

# 7.5 Serious and Unexpected Suspected Adverse Reaction

## (SUSAR)

SUSAR is defined as any significantly untoward medical occurrence, the nature or severity of:

- 1. Which is not consistent with the applicable product information (e.g., Investigator's Brochure) for an unapproved investigational medicinal product.
- 2. Which must be causal relationship with study medication or clinical study.

<sup>†</sup>Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.




## 7.6 SAE Report Procedure

#### 7.6.1 Expedited Reporting of SAEs

Since the clinical study is to be carried out in U.S., when expedited SAEs meet the informed criteria according to the relevant regulations, they will be reported to the Food and Drug Administration (FDA), U.S. by the Sponsor. Written reports should be made on the ADR Reporting Form on Med watch 3500A Form of US FDA, and submitted in a timely fashion according to all relevant regulatory requirements. A copy of this report will also be provided to the principal investigator's local institutional review board if necessary. All SAEs will be monitored until they are resolved or until the principal investigator assesses them as irreversible, chronic, or stable, or until the subject dies. During the clinical trial, if expedited SAEs occur, the investigator should inform the sponsor/CRO within 24 hours by fax and/or telephone.

Principal investigator: Dr. Keith McBurnett

Phone: +1-415-476-7892

Address: 401 Parnassus Ave., Langley Porter Building, San Francisco, California, USA

#### 7.6.2 IRB Notification

Reports of serious adverse events will be communicated to IRB:

- Fatal or life-threatening SUSAR: Should be reported to IRB in the 7 calendar days and detailed written documents should be provided within 15 days after being aware of the event.
- Non-Fatal or life-threatening SUSAR: Should be reported to IRB no later than 15 calendar days.
- Non-SUSAR SAE: Should be reported to IRB following each IRB regulations.

#### 7.6.3 Record Retention

All telephone/fax reports must be followed with a written narrative summary of the adverse event and any sequel. These narratives, which confirm the information collected by telephone and may provide additional information not available at the time of the initial report, must be reviewed by the clinical monitor within seven calendar days following the telephone/fax report to sponsor.




## 8. Statistic Methods

## **8.1 Sample Size Determination**

In part I study, six subjects each will be evaluated for safety and efficacy assessments at 1 and then 2 capsules TID dose for total 56 days (28 days at each dose).

#### 8.2 Statistical Method

Simple descriptive statistics with 95% confidence interval will be performed with data collected in this study wherever applicable. All data shall be tabulated and presented in the study report. The safety and efficacy data will be analyzed using the non-parametric method wherever appropriate.

The purpose for Part I is exploratory in safety and the formal statistical analysis will not be needed. The descriptive statistics will be provided. Safety endpoints will be listed and summarized as appropriate: median and range for continuous data; frequencies, total numbers and percentages for categorical data.

## 8.3 Analysis of Efficacy and Safety

The efficacy measures are conducted on the per-protocol (PP) and intent-to-treat (ITT) basis. The per protocol will be defined as (1) The drug compliance is at least 80%; (2) Subjects have completed data to determine the primary endpoint; (3) Subjects cannot have protocol deviation. The protocol deviation will be defined as (1) Inclusion or exclusion criteria not satisfied; (2) Not permitted concomitant medications. An intent-to-treat (ITT) basis will be defined as the data are analyzed on patients who take at least one dose of study medication and have any post-baseline measurements collected. The safety measures are conducted on the patients who take at least one dose of study medication. The data are analyzed utilizing the last observation carried forward (LOCF) technique to impute the missing data.

The efficacy and safety information recorded on CRF will be summarized by tables presented in frequency and percentage for categorical variables, in mean with SD as well as median with the minimum and maximum for continuous variables. All adverse events

Protocol




will be summarized with coding term, severity, relationship to study drug by frequency tables with the counts and percentage. In addition, serious adverse events will be listed with event narration.

# 8.4 Premature Termination and Handling of Missing Data

Any premature termination of the study therapy will be recorded in CRF. Listing of the subjects with premature termination will be provided with the dates and reasons. Missing data caused by premature termination will be utilized the last observation carried forward (LOCF).




# 9. Quality Control and Quality Assurance

## 9.1 Study Monitoring

The clinical monitor from sponsor-designated contract research organization (CRO) will be responsible for overseeing the progress of a clinical trial to be conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), GCP, and the applicable regulatory requirements. All written informed consent and CRFs will be carefully reviewed and the accuracy of the data will be validated by clinical monitor. During the COVID-19 public health emergency, the monitoring can be performed remotely, but it should be documented.

## 9.2 Sponsor Auditing

Prior to locking the database of safety, the representative of Sponsor's quality assurance department may visit the Investigator's site to implement an audit of study. The audit will to determine the compliance of Investigator with protocol, GCP and applicable regulations. Besides, auditors will assess the accuracy of clinical data record. The Investigator and trial personnel need to cooperate with auditor to facilitate the process of audit.

# 9.3 Inspected by Regulatory Authorities

Local regulatory authority may visit the Investigator to conduct an inspection of this study and the site. The Investigator must make the trial-related records accessible to regulatory agency inspectors. In addition, the Investigator needs to notify the Sponsor immediately when contacted with regulatory authority for the inspection.




#### 10. Ethical Considerations

#### 10.1 Confidential

All information about study subjects will be kept confidential in accordance with the applicable regulatory requirement, to protect and respect the privacy of study subjects. Only the members performed study-related processes, including trial-related monitoring, audits, IRB/IEC review, and regulatory inspection, could directly access to source data/documents.

#### 10.2 Protocol Amendment

Any amendment to the Protocol which deemed necessary as the study progresses will be fully discussed by Investigator and the Sponsor. A written amendment must be submitted to US FDA and Chairman of the IRB, except when the change(s) involves only logistical or administrative aspects of the trial (e.g. change in clinical monitors or change of telephone numbers). Investigator must wait for their approvals of the protocol amendment before implementing the changes. A protocol change intended to eliminate an apparent immediate hazard to trial subjects may be implemented immediately while simultaneously informing FDA /IRB.

When, in the judgment of Chairmen of the IRB, Investigator and/or the Sponsor, the amendment to the Protocol substantially alters the study design and/or increases the potential risk to the subjects, the currently approved written informed consent form will be modified according to the modification. A second informed consent will be obtained from subjects enrolled in the study before further participation.

#### 10.3 Informed Consent

Written informed consent must be reviewed and approved by IRB. Informed consent will be designed to provide detailed information, including explanation of the purpose of this study, the risks and discomforts involved, potential benefits and all basic elements required by regulatory agencies, to participants. Investigator (or his or her qualified designees) will be responsible for explaining the contents of the informed consent to participants as clear as possible. Once it is felt that the subject understands the implications

Protocol




of participating, the written informed consent form shall be signed by the subject and a witness. The written informed consent will be obtained from each subject before any study related procedures (including any pre-treatment procedures) are performed.

## 10.4 Institutional Review Board (IRB)

This study is conducted to be consistent with the principles of the Declaration of Helsinki and GCP. This protocol and any supplementary documents, including written informed consent form, subject recruitment advertisements and Investigator's Brochure, must be reviewed and approved by IRB of the UCSF Medical Center qualified with local legal prescriptions prior to study initiation. The members of IRB are average thirty people, including medical doctors, professors of pharmacology and members whose primary area of interest is in the nonscientific area such as law and social welfare policy. One group of members of IRB meet once a month. Any changes in protocol must be received the IRB approval/favorable opinion in advance of use except for the immediate hazards to trial subjects. Investigator shall submit a status report to IRB at the end of the study. IRB must be notified by the Investigators promptly for all unanticipated problems involving risk to human subjects or others. Investigator is required to maintain an accurate and complete record of all written submissions made to IRB and must agree to share all such documents and reports with the Sponsor and any regulatory agency.




# 11. Data Handling and Record Keeping

An EDC (electronic data capture) system may be used in this study to handle data in an electronic CRF. Follow the EDC system guideline when using it.

# 11.1 Data Handling and Collection

#### 11.1.1 Study Specific Binders

Four types of binder will be utilized in this study:

- Subject Binder: Containing informed consent, all case report forms (not applicable for eCRF) and certain source documents collected for each subject entered the treatment period of the study. Each Subject Binder will have tab dividers for the laboratory printouts. Subject Binders will be kept at each study center.
- Screening Binder: Containing all case report forms of subjects participated in the screening period but found ineligible for entering the treatment period of the study.
   Screening Binders will be kept at each study center
- Generic Forms Binder: Containing enough blank generic case report forms for all subjects participating in the study.
- Study Center File: Documents pertinent to the conduct of this study will be filed in this binder.

#### 11.1.2 Responsibilities of Investigators

Protocol

The Investigator shall process, prepare and maintain complete and accurate study procedure and documentation in compliance with GCP standards and local laws, rules and regulations. It is the Investigators' responsibility to ensure that the designated CRC for this study at the hospital fully understands his/her responsibilities and has the ability to fulfill all the relevant tasks on behalf of the Investigator in many occasions. For each subject enrolled, a CRF must be completed and signed by the Investigator, no matter if this subject has completed the study or not. The Investigator agrees to fully cooperate and assist the clinical monitor in performing their duties, including enabling direct access to the relevant hospital and clinic records. Study documentation will be promptly and fully disclosed to




the Sponsor by the Investigator and also shall be made available at the Investigators' site for inspection, copying, review and audit for a reasonable number of times by representatives of the Sponsor or any regulatory agencies. The Investigator agrees to promptly take any reasonable steps that are requested by the Sponsor as a result of an audit to correct the known error in the study documentation and case report forms. The Investigator shall submit to the Sponsor all original case report forms and all reports required by the Protocol when the clinical study have been completed or terminated.

#### 11.1.3 Responsibilities of Clinical Monitor

Clinical monitor shall frequently inspect the source documents (clinic and hospital subject records) and compare them with the CRF at regular time interval throughout the study, to verify the adherence of study execution to the Protocol and confirm the completeness, consistency and accuracy of the data entered. The monitor will perform source data verification by visually comparison between the entries of the CRF and subjects' records, including informed consent, inclusion/exclusion criteria, key variables, drug administration, adverse experience records and safety variables. Additional monitoring will be required if the error rate is unacceptably high.

#### 11.2 Records Retention

#### 11.2.1 Source Document Retention

Source documents refer to any record pertained to a given subject in the study from which study data is, or could be, obtained or verified. This includes, but not limited to, records, charts, notes and laboratory reports. These records, maintained by the Investigator, shall comply with applicable regulations. At the aspect of ICF keeping, one of the original signed informed consent forms for each participant shall be filed with records kept by the Investigator and the other copy should be given to the subject. Besides, progress notes on each visit to the clinic will be required. The progress note of each visit shall at least contain the date of the visit, a general reference to the procedures completed, general subject status remarks including any significant medical findings, and the signature of the clinician making the entry. In addition, any contact with the subject via telephone or other means that provides significant clinical information, such as adverse events, will also be documented in the progress notes. These will be filed with subject records kept by the Investigator and made available for inspection by authorized personnel.




#### 11.2.2 CRF Retention

All information required by the Protocol will be collected on either CRF or source documents. Essential documents should be retained until the Sponsor informs the Investigator that documents are no longer need to be kept.

#### 11.2.3 Record Maintenance

Regulation requires all investigators participating in clinical trials to maintain detailed clinical data for the duration of one of the following periods, whichever is shortest:

- (1) A period of at least two years following the approval date of an application for a marketing permit in support of which the results of the clinical investigation were submitted, or
- (2) A period of two years after the Sponsor notifies the Investigator that no further application is to be filed with the regulatory authority.

The Investigator will not dispose of any record relevant to this study without informing the Sponsor and providing an opportunity for the Sponsor personnel to collect such record. The Investigator shall take full responsibility for maintaining all documentation related to the conduct of this study, including subject records, research data, and pertinent correspondence. These documents are subject to inspection by the Sponsor and appropriate regulatory authorities.

#### 11.3 Study Center File Management

It will be the responsibility of the clinical monitors/CRC to maintain the study center file. The study center file for this study will contain, but not limited to, the information listed below:

- (1) Investigator Brochure.
- (2) Signed Protocol and Amendments approved by both FDA and IRB.
- (3) Copies of FDA and IRB approval letter for this study.
- (4) Curricula Vitae of Investigator and sub-investigator.
- (5) Other documentation of IRB complied with FDA regulations.
- (6) Copy of Informed Consent Form approved by both FDA and IRB.




- (7) All IRB correspondence (reports to IRB, including reports of all death and adverse experience, annual progress reports, final reports, acknowledgement of receipt of report and actions taken by IRB).
- (8) All IND Efficacy and Safety Reports sent to the Investigator.
- (9) Laboratory certification and/or license.
- (10) All written correspondence with the Sponsor.
- (11) Normal ranges of laboratory value for all laboratory tests required by Protocol.
- (12) CRA monitoring logs.
- (13) Drug Invoices and Drug Dispense/Return Records.




# 12. Publication Plan

Sponsor and Investigator will determine authorship and govern other aspects of the publication process related to this trial. All publications must be approved by the Sponsor prior to publication.

## 13. References

- Robert Riesenberg, Joshua Rosenthal, Leslie Moldauer, Christine Peterson. Results of a proof-of-concept, dose-finding, double-blind, placebo-controlled study of RX-10100 (Serdaxin®) in subjects with major depressive disorder. *Psychopharmacology*. 2012; 221 (4): 601-610.
- 2. Wong DT, Threlkeld PG, Best KL, Bymaster FP. A new inhibitor of norepinephrine uptake devoid of affinity for receptors in rat brain. *J Pharmacol Exp Ther*: 1982 Jul;222(1):61-5.
- 3. Bolden-Watson C, and Richelson E. Blockade by newly-developed antidepressants of biogenic amine uptake into rat brain synaptosomes. *Life Sci.* 1993;52(12):1023-9.
- 4. Sanjay Dube, Mary Anne Della, Prasad Rao, et al. A study of the effects of LY2216684, a selective norepinephrine reuptake inhibitor, in the treatment of major depression. Journal of Psychiatric Research 2010; 44(6): 356-363
- 5. Pliszka SR, McCracken JT, Maas JW. Catecholamines in attention-deficit hyperactivity disorder: current perspectives. *J Am Acad Child Adolesc Psychiatry*. 1996 Mar;35(3):264-72.
- 6. Arnsten AF, Steere JC, Hunt RD. The contribution of alpha 2-noradrenergic mechanisms of prefrontal cortical cognitive function. Potential significance for attention-deficit hyperactivity disorder. *Arch Gen Psychiatry*. 1996 May;53(5):448-55.
- 7. Biederman J, and Spencer T. Attention-deficit/hyperactivity disorder (ADHD) as a noradrenergic disorder. *Biol Psychiatry*. 1999 Nov 1;46(9):1234-42.
- 8. Zhou J. Norepinephrine transporter inhibitors and their therapeutic potential. Drugs Future. 2004; 29(12): 1235-44.
- 9. Davids E, Zhang K, Tarazi FI, Baldessarini RJ. Animal models of attention-deficit hyperactivity disorder. *Brain Res Brain Res Rev.* 2003 Apr;42(1):1-21.
- 10. Prediger RD, Pamplona FA, Fernandes D, Takahashi RN. Caffeine improves spatial learning deficits in an animal model of attention deficit hyperactivity disorder (ADHD)




-- the spontaneously hypertensive rat (SHR). *Int J Neuropsychopharmacol.* 2005 Dec;8(4):583-94. Epub 2005 May 9.

- Allen AJ, Kurlan RM, Gilbert DL, Coffey BJ, Linder SL, et al. Atomoxetine treatment in children and adolescents with ADHD and comorbid tic disorders. *Neurology*. 2005 Dec 27;65(12):1941-9.
- 12. Wilens TE, Haight BR, Horrigan JP, Hudziak JJ, Rosenthal NE, et al. Bupropion XL in adults with attention-deficit/hyperactivity disorder: a randomized, placebocontrolled study. *Biol Psychiatry*. 2005 Apr 1;57(7):793-801.
- Spencer TJ, Adler LA, McGough JJ, Muniz R, Jiang H, Pestreich L. Efficacy and safety of dexmethylphenidate extended-release capsules in adults with attentiondeficit/hyperactivity disorder. *Biol Psychiatry*. 2007 Jun 15;61(12):1380-7. Epub 2006 Nov 29.
- 14. Conners, C. K., Erhardt, D., Sparrow, E. (1999). *Conners' Adult ADHD Rating Scales (CAARS) Technical Manual*. Toronto, ON: Multi-Health Systems.
- 15. George J. DuPaul, Thomas J. Power, Arthur D. (1998). *ADHD Rating Scale-IV: Checklists, Norms, and Clinical Interpretation*.